CLINICAL TRIAL: NCT02716129
Title: Post-cesarean Section Analgesic Potency and Side Effects of Intrathecal Morphine and Nalbuphine
Brief Title: The Effect of Adding Nalbuphine to Intrathecal Morphine on Analgesic Efficacy and Side Effects After Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abdelrady S Ibrahim, MD (Other)
Responsible Party: Sponsor-Investigator, Abdelrady S Ibrahim, MD, Assistant professor of Anesthesia and ICU, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB0000871235
Record Dates: First submitted 2016-03-15; First posted 2016-03-23 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Nalbuphine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Morphine group
  Interventions: Drug: Morphine
- Group 2 (Active Comparator): Morphine plus Nalbuphine group
  Interventions: Drug: Morphine plus Nalbuphine

INTERVENTIONS:
Drug: Morphine — 38 patients of this group will receive 10 mg of 0.5% hyperbaric bupivacaine (Buvanest Spinal 0.5% Heavy) with 0.2 mg morphine (Infumorph - Injection 10 mg/mL) in 0.5 ml volume (total volume 2.5 mL). Patients will be preloaded with 10 ml/kg Ringer's lactate solution intravenous.
  Other Names: Infumorph
  Arms: Group 1
Drug: Morphine plus Nalbuphine — 39 patients of this group will receive 10 mg of 0.5% hyperbaric bupivacaine (Buvanest Spinal 0.5% Heavy) with 0.5 mg morphine (Infumorph - Injection 10 mg/mL) plus 0.2 mg nalbuphine (NALUFIN 20MG/ML AMP) in 0.5 ml volume (total volume 2.5 mL). Patients will be preloaded with 10 ml/kg Ringer's lactate solution intravenous.
  Other Names: Infumorph and NALUFIN
  Arms: Group 2

SUMMARY:
The primary endpoint of this study is to investigate the effect of adding nalbuphine to intrathecal morphine on quality of postoperative analgesia and Morphine related side effects post- cesarean delivery.

DETAILED DESCRIPTION:
The study will be performed in Assiut University Hospitals, after obtaining approval from the local ethics committee and written informed patient consent. All patients will have a peripheral IV cannula 18 G inserted; standard non-invasive monitors will be applied. All the patients will be preloaded with 10 ml/kg Ringer's lactate solution intravenous. Intrathecal block under strict aseptic conditions will be performed in sitting position at L3-4 or L4-5 inter-spinous space with 25G pencil-point spinal needle. All patients will receive intrathecal 10 mg of 0.5% hyperbaric bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* age between 16 to 40 years
* ASA physical status I - II

Exclusion Criteria:

* Infection at the site of injection.
* Coagulopathy or other bleeding diathesis.
* Preexisting neurologic deficits.
* History of hypersensitivity to any of the given the drugs.
* Inability to communicate with the investigator and the hospital staff.
* History of chronic opioid us

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours
  Visual Analogue Score

SECONDARY OUTCOMES:
Incidence of postoperative itching | 24 hours
  Visual Analogue Score
number of participants with incidence of postoperative nausea | 24 hours
  Patients number
number of participants with incidence of postoperative vomiting | 24 hours
  Patients number
number of participants with incidence of postoperative postdural puncture headache | 24 hours
  Patients number
number of participants with incidence of postoperative respiratory depression | 24 hours
  Patients number

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrady S Ibrahim, MD, Principal Investigator — Assistant professor of anesthesia and intensive care
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Culebras X, Gaggero G, Zatloukal J, Kern C, Marti RA. Advantages of intrathecal nalbuphine, compared with intrathecal morphine, after cesarean delivery: an evaluation of postoperative analgesia and adverse effects. Anesth Analg. 2000 Sep;91(3):601-5. doi: 10.1097/00000539-200009000-00019. PMID 10960384